CLINICAL TRIAL: NCT06941194
Title: Preventive Application of Single-use Negative Pressure Wound Therapy (sNPWT) in the Postoperative Course of Radiotreatated Limb Sarcoma Surgery a Randomized Clinical Trial
Brief Title: Preventive Application of Single-use Negative Pressure Wound Therapy (sNPWT) in the Postoperative Course of Radiotreatated Limb Sarcoma Surgery
Acronym: PRALISS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Oncologico Veneto IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IOV-SA-01-2024-PRALISS
Record Dates: First submitted 2025-04-16; First posted 2025-04-23 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Sarcoma; Sarcoma,Soft Tissue
Keywords: sarcoma; limbs; high-grade (grade III) soft tissue sarcoma; PICO14
MeSH Terms: conditions — Sarcoma; Lymphoma, Follicular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PICO14 (Experimental): PICO14 is a dressing designed to allow uniform distribution of negative pressure over the surface of a closed surgical incision and is classified as a Class IIb medical device according to Medical Device Directive 93/42/EEC and s.a.u. PICO14 (trade name) has been granted the CE marking in 1994 according to the Medical Device Directive 93/42/EEC and s.a.u.
  It is a portable device, without collection canister, consisting of a sterile pump connected to a multilayer adhesive dressing. The pump is powered by two batteries which provide the continuous negative pressure. The PICO 14 dual dressing kit is intended to be used for up to 14 days on low to moderately exuding wounds.
  Interventions: Device: PICO 14
- Control (No Intervention): patient receive only standard therapy

INTERVENTIONS:
Device: PICO 14 — PICO 14 application after neoadjuvant radiotherapy followed by surgery
  Arms: PICO14

SUMMARY:
Patients will be recruited at the time of the pre-admission visit. During the screening visit the patient will undergo a physical examination and his medical history will be collected. Oncological history and tumor characteristics will be considered and CT-scan imaging will be analysed. ECOG performance status will be reported. If inclusion criteria are respected, the patient will be randomized. The application of the PICO14 study device or standard dressing (dry gauze and plaster) will then be carried out on the day of surgery. For subjects randomized to the treatment arm (Arm A), dressing change with the application of the new PICO14 will occur at day 4+1, day 8±1, and day 14±2. For subjects randomized to the control arm (Arm B), the standard dressing with gauze and plaster is applied. Regardless of the randomization arm the wound assessment via ASEPSIS score will occur at day 4+1, 8±1 and 14±2. During FUP, the dressing can be changed autonomously by the patient if necessary. The information will be recorded on the occasion of the next visit or an extraordinary visit. On day 21, sutures will be removed.

On day 30±2, the total ASEPSIS score will be calculated, in order to evaluate the wound healing.

From day 14±2, regardless of the randomization arm all patients will be treated with standard dressing.

Follow-up visits can be scheduled up to 90 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age
* diagnosis of primary high-grade (grade III) soft tissue sarcoma of the limbs (confirmed histopathologically)
* performed neoadjuvant radiotherapy (short or long-term)
* candidates for wide radical excision surgery
* negative CT scan staging for distant metastasis
* Signing of Informed consent

Exclusion Criteria:

* diagnosis of benign neoplasm
* diagnosis of retroperitoneal or trunk sarcomas;
* candidates to hindquarter or forequarter amputation surgery;
* incomplete wide excision;
* vascular resection;
* other loco-regional treatments (e.g. isolated limb perfusion or electrochemotherapy).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Primary objective and endpoint | Through study completion, an average of 2 years
  Assess, in patients with wide excision surgery of radio treated limb sarcoma, if the preventive application of single-use negative pressure wound dressing (PICO 14) may reduce the incidence of wound complications at 30° day compared to the standard procedure currently in use. Primary objective will be evaluated according to the ASEPSIS score. For each patient the Daily ASEPSIS score will be calculated at days 4, 8 and 14 after surgery.

SECONDARY OUTCOMES:
Secondary objective and endpoint | Through study completion, an average of 2 years
  Evaluate and compare the incidence of long-term wound complications. All complications occurred between day 31 and day 90 after surgery will be collected and reported at the time of appearance, by ASEPSIS score
Third objective and endpoint | Through study completion, an average of 2 years
  Verify the impact of the type of wound dressing in the length of hospital-stay. 2. The length of hospital stay will be calculated as the difference between the date of hospital discharge and the date of surgery
Fourth objective and endpoint | Through study completion, an average of 2 years
  Evaluate the outpatient care time. 3. Outpatient care time will be calculated as the difference between the date of the last outpatient medication and the date of discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Oncologico Veneto, Padua, Italy/Padova, Italy

IPD SHARING:
Plan to Share IPD: Undecided